CLINICAL TRIAL: NCT01498536
Title: Fit for the Fight: Effect of a Multidisciplinary Diet and Exercise Program on Body Weight, Quality of Life and Inflammation in Survivors of Triple-negative Breast Cancer
Brief Title: Effect of Diet and Exercise in Breast Cancer Survivors
Acronym: F4F tri neg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Anne Swisher, Associate Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-22426
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer; Obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: aerobic exercise — 3 times per week for 12-weeks

SUMMARY:
This study seeks to see if a 12-week diet and exercise program improves exercise ability, energy level, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ER/PR/HER2neu negative breast cancer
* at least 3 months after end of treatment
* BMI at least 25

Exclusion Criteria:

* stage IV cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 weeks
  aim for loss of 10% of BMI
quality of life | 12 weeks
  Fatigue, disease-specific symptoms, depression and energy level all assessed by standardized questionnaires

SECONDARY OUTCOMES:
markers of inflammation | 12 weeks
  blood draws at beginning and end of study to analyze any effect on inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States